CLINICAL TRIAL: NCT04224610
Title: The Utility of (Fractional Flow Reserve)FFR Before and After Successful Percutaneous Coronary Intervention
Status: Active, not recruiting | Type: Observational
Sponsor: Central Arkansas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 779601
Record Dates: First submitted 2019-08-12; First posted 2020-01-13 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to analyze the data of patients who underwent FFR evaluation at CAVHS to evaluate the impact of PCI on coronary hemodynamics in patients with baseline ischemic FFR, the potential etiologies of suboptimal FFR post PCI, determine potential measures taken to correct persistently suboptimal FFR and PCI, and determine rate of clinical events, utility of routine Post PCI FFR strategy compared to pre PCI FFR strategy only, and evaluate the "Warranty Period" of non-ischemic FFR in different sub groups.

DETAILED DESCRIPTION:
Background Fractional flow reserve (FFR) measurement has become the gold standard for establishing ischemia in the intermediate lesion detected at angiography. As such, it is a Class IA indication in the European Guidelines and IIA in the ACC/AHA Guidelines. Furthermore, an FFR guided strategy for selecting percutaneous revascularization has been shown in multiple randomized trials and numerous large registries to confer favorable long term clinical outcomes. Importantly, the cost effectiveness and the consequent efficient resource utilization of an FFR guided approach have been rigorously established. Despite this solid evidence base, data from the National Cardiovascular Data Registry (NCDR ®) NCDR CathPCI Registry evaluating current practice (2009-2010) in >61000 patients with intermediate coronary stenosis (40-70%) undergoing PCI showed that only 6.1% patients underwent FFR evaluation while 20% underwent intravascular ultrasound (IVUS) evaluation; the majority of intermediate lesions underwent percutaneous coronary intervention (PCI) based on coronary angiography alone.

While it has been shown that "deferring PCI" for FFR >0.80 is safe, factors affecting the negative predictive value of FFR and hence the prognostic utility are not fully elucidated. The biology of disease is not the same in all patients as was shown by a recent meta-analysis which found that FFR threshold for intervention was influenced by factors such as the presence of left main disease and diabetes . In the light of this information it is conceivable that the warranty period of any given value of non-ischemic FFR will differ in patients with and without such factors. The concept is not new and has previously been applied to myocardial perfusion imaging (MPI) where it was determined that the warranty period for event free survival after a negative MPI was lower in those with diabetes and CKD.

Despite the robust efficacy of PCI in relieving angina, a substantial proportion of patients continue to experience clinical events including death, myocardial infarction, or recurrent angina necessitating repeat revascularization; even in the drug eluting stent (DES) era. Accumulating evidence over the past 15 years has shown that as much as angiographic evaluation is significantly limited in assessing lesion severity, likewise angiographic evaluation of PCI results is also severely limited. Data from FFR, optical coherence tomography (OCT) and IVUS based studies have shown that based on angiography alone, a significant proportion of patients undergoing PCI and stenting have suboptimal results which in turn translate into downstream adverse outcomes. Whereas FFR has been shown to determine the hemodynamic significance of a coronary stenosis and FFR guided PCI proven to significantly improve clinical outcomes, a significant proportion of patients even in the FFR guided PCI group continue to experience significant events. For instance, in the pivotal FAME trial, the one year major adverse cardiac events (MACE) event rate was 13.2% in the FFR guided PCI arm (albeit 30% lower than the angiographically guided PCI group) and 20% at 2 years.

Multiple factors including stent under expansion/ malapposition, geographic miss of the culprit lesion or placement in diseased bed, diffuse atherosclerosis are not frequently missed on angiography. In this context, the utility of FFR for assessing the "effectiveness of PCI" has emerged as an attractive strategy. Studies dating back to 1999, have demonstrated the robust utility of post PCI FFR in evaluating the efficacy of PCI. Post PCI FFR has been shown to correlate with optimal stenting and PTCA as determined by IVUS. Additionally, post PCI FFR has been shown to be a predictor of major adverse events including death, myocardial infarction (MI), and target vessel revascularization (TVR).

Methods This project will be a retrospective chart review of all consecutive patients who have undergone FFR evaluation at the CAVHS between 3/2009 till 3/2015. Demographic data (age and gender), risk factor profile, clinical presentation , baseline lab data, ejection fraction (EF) will be retrieved from the VA CPRS system. Details of coronary angiography including number of diseased vessels, pre and post stenosis (% luminal diameter), stent number, type and size will be recorded. Additional variables related to the PCI will be recorded as shown below and attached Excel sheet.

Follow up and Clinical endpoints This is a RETROSPECTIVE CHART REVIEW. All follow up information and clinical endpoints will be collected from CPRS. There will be NO DIRECT PATIENT CONTACT. In-hospital events will include major adverse events, such as Q wave myocardial infarction (MI), need for emergency surgery, or death during hospitalization. Clinical outcomes including death, myocardial infarction, instent restenosis (ISR) and target vessel revascularization.) will be recorded at 30 days and at last follow up (retrieved from CPRS). This information will be retrieved from inpatient and outpatient electronic records for patients (CPRS).

Statistical Analysis Comparison of baseline, angiographic, procedural and outcome variables for patients with FFR>0.9 and <0.9 will be done using unpaired Student's t-test for continuous variables and the chi square test( χ2 ) for categorical or dichotomous variables. Unadjusted annual event rates for those with and without FFR>0.9 will be calculated by first estimating overall event rates for these groups through calculation of Kaplan-Meier(K-M) curves, then dividing the event rate by the mean follow-up time for each of the groups. Additionally, median pre and post FFR, (%) diameter stenosis will be calculated for patients with and without clinical outcomes.

Univariate predictors of post PCI, FFR,and MACE will recorded. Multivariate stepwise logistic regression analysis will be applied to identify independent predictors (adjusted OR with 95% CI) for a) Post PCI FFR>0.9 and b) MACE.

Receiver operator curve analysis will be performed to assess the optimal "cutoff" value of post PCI FFR for predicting MACE in our population.

The level of statistical significance will be a priori set at <0.05, and a 2-sided probability value used for the analyses. All statistical calculations will be performed using MedCalc Statistical Software.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have undergone FFR at CAVHS between 3/2009 and 3/2015.

Exclusion Criteria:

* No FFR

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have undergone FFR at CAVHS between 3/2009 and 3/2015 will be reviewed. Comparison of baseline, angiographic, procedural and outcome variables for patients with FFR>0.9 and <0.9 will be done using unpaired Student's t-test for continuous variables and the chi square test( χ2 ) for categorical or dichotomous variables. Unadjusted annual event rates for those with and without FFR>0.9 will be calculated by first estimating overall event rates for these groups through calculation of Kaplan-Meier(K-M) curves, then dividing the event rate by the mean follow-up time for each of the groups. Additionally, median pre and post FFR, (%) diameter stenosis will be calculated for patients with and without clinical outcomes.Univariate predictors of post PCI, FFR,and MACE will recorded.
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2009-03-01 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact of PCI | Immediately post procedure
  • Evaluate the impact of PCI on coronary hemodynamics in patients with baseline ischemic FFR compared to final FFR

SECONDARY OUTCOMES:
Potential etiologies of suboptimal FFR | Immediately post procedure
  • Evaluate potential etiologies of suboptimal FFR post PCI (Identify clinical, angiographic and IVUS/OCT predictors of normalized (FFR>0.96), optimal (FFR>0.85) and suboptimal hemodynamics (<0.8-0.85
Determine potential corrective measures | Immediately post procedure
  • Determine potential measures taken to correct persistently suboptimal FFR post PCI including additional stenting; IVUS/OCT evaluation; post dilation
Determine rate of clinical events | Immediately post procedure
  • Determine potential measures taken to correct persistently suboptimal FFR post PCI including additional stenting; IVUS/OCT evaluation; post dilation
Compare post PCI FFR strategy to pre PCI FFR only | Immediately post procedure
  • Evaluate the utility of routine Post PCI FFR strategy to compare final FFR value to pre PCI FFR only strategy in different patient subsets including those with stable angina, ACS (Unstable angina/NSTEMI).
Evaluate "Warranty Period" | Through end of study, approximately 5 years
  • Evaluate the "Warranty Period" (period of no clinical events) of non-ischemic FFR in different sub groups (diabetes, hypertension, chronic kidney disease ).

CONTACTS AND LOCATIONS:
Overall Officials: Barry Uretsky, MD, Principal Investigator — CAVHS

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lotfi A, Jeremias A, Fearon WF, Feldman MD, Mehran R, Messenger JC, Grines CL, Dean LS, Kern MJ, Klein LW; Society of Cardiovascular Angiography and Interventions. Expert consensus statement on the use of fractional flow reserve, intravascular ultrasound, and optical coherence tomography: a consensus statement of the Society of Cardiovascular Angiography and Interventions. Catheter Cardiovasc Interv. 2014 Mar 1;83(4):509-18. doi: 10.1002/ccd.25222. Epub 2013 Nov 13. No abstract available. PMID 24227282
- [Background] Hanekamp CE, Koolen JJ, Pijls NH, Michels HR, Bonnier HJ. Comparison of quantitative coronary angiography, intravascular ultrasound, and coronary pressure measurement to assess optimum stent deployment. Circulation. 1999 Mar 2;99(8):1015-21. doi: 10.1161/01.cir.99.8.1015. PMID 10051294
- [Background] Pijls NH, Klauss V, Siebert U, Powers E, Takazawa K, Fearon WF, Escaned J, Tsurumi Y, Akasaka T, Samady H, De Bruyne B; Fractional Flow Reserve (FFR) Post-Stent Registry Investigators. Coronary pressure measurement after stenting predicts adverse events at follow-up: a multicenter registry. Circulation. 2002 Jun 25;105(25):2950-4. doi: 10.1161/01.cir.0000020547.92091.76. PMID 12081986
- [Background] Fearon WF, Luna J, Samady H, Powers ER, Feldman T, Dib N, Tuzcu EM, Cleman MW, Chou TM, Cohen DJ, Ragosta M, Takagi A, Jeremias A, Fitzgerald PJ, Yeung AC, Kern MJ, Yock PG. Fractional flow reserve compared with intravascular ultrasound guidance for optimizing stent deployment. Circulation. 2001 Oct 16;104(16):1917-22. doi: 10.1161/hc4101.097539. PMID 11602494
- [Background] Bech GJ, Pijls NH, De Bruyne B, Peels KH, Michels HR, Bonnier HJ, Koolen JJ. Usefulness of fractional flow reserve to predict clinical outcome after balloon angioplasty. Circulation. 1999 Feb 23;99(7):883-8. doi: 10.1161/01.cir.99.7.883. PMID 10027810
- [Background] Klauss V, Erdin P, Rieber J, Leibig M, Stempfle HU, Konig A, Baylacher M, Theisen K, Haufe MC, Sroczynski G, Schiele T, Siebert U. Fractional flow reserve for the prediction of cardiac events after coronary stent implantation: results of a multivariate analysis. Heart. 2005 Feb;91(2):203-6. doi: 10.1136/hrt.2003.027797. PMID 15657233
- [Background] Leesar MA, Satran A, Yalamanchili V, Helmy T, Abdul-Waheed M, Wongpraparut N. The impact of fractional flow reserve measurement on clinical outcomes after transradial coronary stenting. EuroIntervention. 2011 Dec;7(8):917-23. doi: 10.4244/EIJV7I8A145. PMID 22157476
- [Background] Dupouy P, Gilard M, Morelle JF, Furber A, Aptecar E, Cazaux P, Slama M, Feldman LJ, Wittenberg O, Pernes JM, Huret B, Commeau P, Boschat J, Teiger E, Lafont A, Steg PG, Dubois Rande JL. Usefulness and clinical impact of a fractional flow reserve and angiographic targeted strategy for coronary artery stenting: FROST III, a multicenter prospective registry. EuroIntervention. 2005 May;1(1):85-92. PMID 19758882